CLINICAL TRIAL: NCT02084862
Title: Ultrasound Guided Percutaneous Tracheostomy Compared to Bronchoscopy Guided Percutaneous Tracheostomy - A Randomized Non-inferiority Trial
Brief Title: Ultrasound Guided Percutaneous Tracheostomy Compared to Bronchoscopy Guided Percutaneous Tracheostomy
Acronym: TRACHUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luiz Marcelo Sá Malbouisson, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11410; 488506 (Other: CAPPesq)
Record Dates: First submitted 2014-02-05; First posted 2014-03-12 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Tracheostomy Complications
Keywords: Tracheostomy; Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Ultrasound guided percutaneous tracheostomy
  Interventions: Device: Ultrasound guided percutaneous tracheostomy
- Bronchoscopy (Active Comparator): Bronchoscopy guided percutaneous tracheostomy
  Interventions: Device: Bronchoscopy guided percutaneous tracheostomy

INTERVENTIONS:
Device: Ultrasound guided percutaneous tracheostomy — Ultrasound guided percutaneous tracheostomy
  Arms: Ultrasound
Device: Bronchoscopy guided percutaneous tracheostomy — Bronchoscopy guided percutaneous tracheostomy
  Arms: Bronchoscopy

SUMMARY:
TRACHUS trial is a randomized non-inferiority trial designed to evaluate the safety and efficacy of ultrasound guided percutaneous tracheostomy compared to bronchoscopy guided percutaneous tracheostomy.

DETAILED DESCRIPTION:
TRACHUS trial is a randomized non-inferiority trial designed to evaluate the safety and efficacy of ultrasound guided percutaneous tracheostomy compared to bronchoscopy guided percutaneous tracheostomy.

Patients will be randomly assigned to be submitted to ultrasound or bronchoscopy guided percutaneous tracheostomy and then the procedure related complications and clinical outcomes will be evaluated and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* All intubated and mechanically ventilated patients indicated for a tracheostomy by the ICU assistant team

Exclusion Criteria:

* Patients with unfavorable anatomy judged by the patient assistant team (short neck, tracheal deviation, cervical anatomical anomaly, previous cervical surgery, cervical trauma or inability to perform neck extension), preference for surgical tracheostomy by the patient assistant team or patients unable to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Procedure failure | During PDT - an expected average of 15 minutes
  Combined endpoint procedure failure (defined as conversion to surgical tracheostomy, or associated use of bronchoscopy in the case of ultrasound-guided tracheostomy or associated use of ultrasound in bronchoscopy-guided tracheostomy) or occurrence of of a major complications defined as transfusion, hypotension or surgical intervention in the operative room due to bleeding, tracheal laceration, tracheal posterior wall injury, esophageal injury, tracheoesophageal fistula, cardiorespiratory arrest or death due to tracheostomy.

SECONDARY OUTCOMES:
Hypoxemia | During PDT - an expected average of 15 minutes
  Drop in peripheral oxygen saturation < 90% for more than 2 minutes as measured by pulse oxymeter during the procedure
Hypotension | During PDT - an expected average of 15 minutes
  Systolic blood pressure < 90mmHg for more than 5 minutes and any intervention aimed to raise blood pressure such as vasopressor or fluid administration.
Pneumothorax | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Pneumothorax due to the PDT detected by clinical examination during the procedure or chest x-ray after the procedure.
Atelectasis | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Atelectasis due to the PDT detected by clinical examination during the procedure or chest x-ray after the procedure.
Conversion to surgical tracheostomy | During PDT - an expected average of 15 minutes
  Conversion to surgical tracheostomy due to technical limitations or complications during PDT.
Tracheal posterior wall injury | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Tracheal posterior wall injury as detected by bronchoscopy after the procedure
Accidental decanulation | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Accidental decanulation after the procedure during Hospital stay
Cardiorespiratoty arrest | During PDT - an expected average of 15 minutes
  Cardiorespiratory arrest due to PDT
Death | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Death due to PDT complications
Liberation from mechanical ventilation | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Breathing without ventilator assistance for at least 48 hours after the PDT
Length of ICU Stay | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Length of ICU Stay
Length of Hospital Stay | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Length of Hospital Stay
Length of Mechanical Ventilation | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Length of Mechanical Ventilation
Surgical site infection | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Surgical site infection defined as antibiotic introduction directed to surgical site
Tracheal ring fracture | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Tracheal ring fracture detected by bronchosocopy after the PDT
Tracheal-esophageal fistula | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Trachealesophageal fistula detected by bronchosocopy after PDT
Minor bleeding | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Clinical relevant bleeding attributed to PDT defined as need for any intervention to stop the bleeding such as vessel ligature or local wound care.
Major bleeding | During the procedure - an expected average of 15 minutes
  Blood transfusion or hypotension or surgical intervention in the operating room due to bleeding during PDT
Major bleeding | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Blood transfusion or hypotension or surgical intervention in the operating room due to bleeding related to PDT during hospital stay after the procedure

OTHER OUTCOMES:
Procedure duration | During PDT - an expected average of 15 minutes
  Time elapsed between skin incision and connection of mechanical ventilation to tracheostomy cannula
Time to procedure performance | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Time elapsed between participant randomization and PDT performance

CONTACTS AND LOCATIONS:
Overall Officials: André Gobatto, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Cínicas da Universidade de São Paulo, São Paulo, São Paulo, Brazil